CLINICAL TRIAL: NCT04057612
Title: Correlation Between Core Temperature and Skin Temperature Near Carotid Artery Measured by 3M™ Bair Hugger™ in Pediatrics
Brief Title: Correlation Between Core Temperature and Skin Temperature in Pediatrics
Acronym: temperature
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical Assistant Professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-19-277
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Temperature Change, Body; Anesthesia; Children, Only
Keywords: pediatric; temperature; general anesthesia
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric participants: Participants' temperature measured at 2 places at the same time
  * Esophagus
  * Skin near to carotid artery
  Interventions: Other: Esophagus temperature monitoring; Other: Carotid artery temperature monitoring

INTERVENTIONS:
Other: Esophagus temperature monitoring — Measuring core temperature by esophageal stethoscope
  Other Names: core temperature
Other: Carotid artery temperature monitoring — Measuring temperature on skin near to carotid artery using 3M™ Bair Hugger™ temperature monitoring system
  Other Names: 3M™ Bair Hugger™ temperature monitoring

SUMMARY:
During general anesthesia, temperature monitoring is critical especially in pediatrics. Recently developed 3M™ Bair Hugger™ skin temperature which is applied on temporal artery is correlated with core temperature measure by esophageal prove in several studies. Conventional skin temperature over carotid artery is also correlated with core temperature in several studies. The purpose of this study is comparing 2 methods of temperature monitoring in pediatrics. First, conventional core temperature measure by esophageal stethoscope. Second, 3M™ Bair Hugger™ applying on carotid artery.

DETAILED DESCRIPTION:
Core temperature should be monitored under general anesthesia. Because patients are prone to hypothermia during surgery, besides, pediatric patients are more vulnerable in temperature control. Conventional core temperature is monitored at esophagus, rectum, nasopharynx. But some of them are invasive and impossible in sometimes. Recently developed 3M™ Bair Hugger™ skin temperature which is applied on temporal artery is correlated with core temperature measured by esophageal prove in several studies. Its mechanism is making zero heat flux on skin applied. But it also cannot apply in head or facial surgery. Other studies showed conventional skin temperature over carotid artery is also correlated with core temperature. The investigators hypothesized using 3M™ Bair Hugger™ on carotid artery could be alternative method measuring core temperature. The purpose of this study is comparing 2 methods of temperature monitoring in pediatrics. First, conventional core temperature measure by esophageal stethoscope. Second, 3M™ Bair Hugger™ applying on carotid artery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled operation under general anesthesia
* Who need esophageal temperature monitoring
* American society of anesthesiology physical status 1 or 2

Exclusion Criteria:

* Body mass index > 35 kg/m2
* Who cannot be inserted esophageal temperature prove
* Patients with fever > 38'C
* History of malignant hyperthermia

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 1 to 5 years old who scheduled surgery under general anesthesia. Who need esophageal temperature monitoring for routine monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Esophageal core temperature measured by stethoscope, ℃ | 3 hours (during general anesthesia)
  Temperature measured by esophageal stethoscope, ℃
Carotid skin temperature by 3M™ Bair Hugger™, ℃ | 3 hours (during general anesthesia)
  Temperature measured by 3M™ Bair Hugger™ near to carotid artery, ℃

SECONDARY OUTCOMES:
Room temperature, ℃ | 3 hours (during general anesthesia)
  Operating room temperature, ℃

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided